CLINICAL TRIAL: NCT07333456
Title: The Effects of Vibration on Lower Limb Muscle Strength, Functional Status, and Psychological Health in Stroke Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tri-Service General Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Yu-Jung Tseng, Principal Investigator, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: YJTseng; NSTC 112-2314-B-016-069 (Other Grant/Funding Number: Ministry of Science and Technology); C202305047 (Other: Institutional Review Board of Tri-Service General Hospital, National Defense Medical Center); C202105050 (Other: Institutional Review Board of Tri-Service General Hospital, National Defense Medical Center)
Record Dates: First submitted 2025-09-29; First posted 2026-01-12 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Stroke
Keywords: stroke; early rehabilitation; vibration; Lower limb muscle strength; Functional status; Psychological health
MeSH Terms: conditions — Stroke; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Active Comparator): Receives only standard stroke treatment and rehabilitation therapy.
  Interventions: Behavioral: regular treatment
- Stationary cycling training (Experimental): In addition to standard stroke treatment, participants receive 5 days of stationary cycling training in the acute stroke unit beginning 1-2 days after admission (at least 24 hours after the stroke onset). The cycling session lasts approximately 30 minutes, including a 5-minute warm-up, 20-minute training session, and 5-minute cool-down.
  Interventions: Behavioral: early rehabilitation; Behavioral: regular treatment
- Stationary cycling training combined with localized vibration therapy (Experimental): In addition to standard rehabilitation, participants receive 5 days of stationary cycling training combined with localized vibration therapy administered using a wearable vibration device. Vibration parameters are set at a frequency of 30 Hz and amplitude of 1 mm, targeting the lower-leg muscle groups. Each session lasts 30 minutes and begins within 1-2 days of admission.
  Interventions: Behavioral: wearable vibration; Behavioral: early rehabilitation; Behavioral: regular treatment
- Stationary cycling training combined with vertical vibration therapy (Experimental): In addition to standard rehabilitation, participants receive 5 days of stationary cycling training combined with vertical vibration therapy for the lower limbs. Vibration parameters are set at a frequency of 20 Hz and amplitude of 3 mm. Each session also lasts 30 minutes and begins within 1-2 days of admission.
  Interventions: Behavioral: vertical vibration; Behavioral: early rehabilitation; Behavioral: regular treatment

INTERVENTIONS:
Behavioral: wearable vibration — In addition to standard rehabilitation, participants receive 5 days of stationary cycling training combined with localized vibration therapy administered using a wearable vibration device. Vibration parameters are set at a frequency of 30 Hz and amplitude of 1 mm, targeting the lower-leg muscle groups. Each session lasts 30 minutes and begins within 1-2 days of admission.
  Other Names: early rehabilitation
  Arms: Stationary cycling training combined with localized vibration therapy
Behavioral: vertical vibration — In addition to standard rehabilitation, participants receive 5 days of stationary cycling training combined with vertical vibration therapy for the lower limbs. Vibration parameters are set at a frequency of 20 Hz and amplitude of 3 mm. Each session also lasts 30 minutes and begins within 1-2 days of admission.
  Other Names: early rehabilitation
  Arms: Stationary cycling training combined with vertical vibration therapy
Behavioral: early rehabilitation — In addition to standard stroke treatment, participants receive 5 days of stationary cycling training in the acute stroke unit beginning 1-2 days after admission (at least 24 hours after the stroke onset). The cycling session lasts approximately 30 minutes, including a 5-minute warm-up, 20-minute training session, and 5-minute cool-down.
  Arms: Stationary cycling training; Stationary cycling training combined with localized vibration therapy; Stationary cycling training combined with vertical vibration therapy
Behavioral: regular treatment — Receives only standard stroke treatment and rehabilitation therapy.

SUMMARY:
The goal of this clinical trial is to the effect of vibration training on lower limb muscle strength, functional status and psychological health of stroke patients. The main questions it aims to answer are:

* Lower limb muscle strength was measured using the Medical Research Council Manual Strength Test.
* Functional status was measured using Postural Assessment Scale for Stroke, and the Barthel scale.
* Psychological health was measured using the Hospital Anxiety and Depression Scale.

Participants will be randomly assigned to four groups:

1. Control group: Receives only rehabilitation training and standard treatment.
2. Comparison group: Receives rehabilitation training, standard treatment, and a 30-minute stationary cycling intervention during hospitalization for 5 days.
3. Experimental group 1: Receives rehabilitation training, standard treatment, and a 30-minute wearable lower-limb high-frequency, low-amplitude vibration therapy during hospitalization for 5 days, followed by 30 minutes of stationary cycling.
4. Experimental group 2: Receives rehabilitation training, standard treatment, and a 30-minute vertical lower-limb low-frequency, high-amplitude vibration therapy during hospitalization for 5 days, followed by 30 minutes of stationary cycling.

All participants will undergo an initial measurement within 4 hours of admission, followed by the second and third measurements after the 5-day intervention and on the day of discharge, respectively.

DETAILED DESCRIPTION:
Standard care for all study participants includes conventional rehabilitation therapy for stroke. This therapy involves physical therapy (e.g., posture training, endurance training, muscle strength training) and occupational therapy provided at the rehabilitation center. Such rehabilitation typically begins 3-6 days after admission and is administered by a physical or occupational therapist.

* Control group: Receives only standard stroke treatment and rehabilitation therapy.
* Comparison group: Additionally, using stationary lower leg pedal bike (WP-698) with moderate intensity.
* Experimental group 1: In addition to standard rehabilitation, participants receive 5 days of stationary cycling training combined with localized vibration therapy with a wearable vibration device (Myovolt).
* Experimental group 2: In addition to standard rehabilitation, participants receive 5 days of stationary cycling training combined with vertical vibration therapy for the lower limbs with COZY FIT vertical vibration machine (HY-806-BK)

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized with a diagnosis of acute ischemic stroke (cerebral infarction).
2. Stroke onset occurred within three days of admission.
3. Age between 20 and 80 years old.
4. Ability to communicate verbally or non-verbally and understand Mandarin or Taiwanese.
5. Normal cognitive function (MMSE ≥ 21).
6. Disability level assessed as 1-4 on the modified Rankin Scale (mRS)
7. Willingness to participate in the study and agree to random group allocation.

Exclusion Criteria:

1. Diagnosed with transient ischemic attack (TIA) accompanied by vision or hearing impairments.
2. Disability level of mRS ≥ 5 (severe disability requiring bedridden care).
3. Acute or chronic neurological or musculoskeletal injuries in the lower limbs or history of joint surgery within the past six months.
4. Presence of a pacemaker.
5. Unstable or significant cardiovascular or cardiac disease, cancer history, end-stage renal disease requiring hemodialysis, or diagnosed psychiatric disorders, especially depression.
6. Patients transferred from other hospital wards or intensive care units.
7. Hospitalization exceeding 21 days due to other medical or surgical conditions (e.g., infections) or hospitalization shortened to fewer than seven days due to hospital transfers or seeking alternative therapies.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2025-04-26 (Actual); Study Completion 2025-04-26 (Actual)

PRIMARY OUTCOMES:
Lower-limb muscle strength | All participants will undergo an initial measurement within 4 hours of admission, followed by the second and third measurements after the 5-day intervention and on the day of discharge, an average of 11 days , respectively.
  Using the Medical Research Council Manual Strength Test. Muscle strength was assessed by evaluating the ability of the limbs to move against gravity or applied resistance, using a grading scale ranging from 0 to 5. Higher scores indicate better muscle strength. A score of 0 indicates no visible or palpable muscle contraction; 1 indicates only visible or palpable muscle contraction; 2 indicates joint movement with gravity eliminated; 3 indicates observable joint movement against gravity but not against resistance; 4 indicates joint movement against gravity with some resistance; and 5 indicates joint movement with full resistance against both gravity and applied resistance.
Functional status | All participants will undergo an initial measurement within 4 hours of admission, followed by the second and third measurements after the 5-day intervention and on the day of discharge, an average of 11 days, respectively.
  Using Postural Assessment Scale for Stroke, and the Barthel scale. The scale consists of 12 items and is scored using a four-point scale (0-1-2-3), with a total score ranging from 0 to 36. Higher scores indicate better postural control and balance function. It primarily assesses two domains: (1) stability of body posture, including static and dynamic balance, and (2) the ability to change body positions, encompa Barthel scale: The scale primarily assesses activities of daily living, including feeding, grooming, toileting, bathing, dressing, bowel and bladder control, transfers between a wheelchair and bed, walking on a level surface or wheelchair propulsion, and stair climbing. The total score ranges from 0 to 100. Scores of 0-20 indicate complete dependence, 21-60 indicate severe dependence, 61-90 indicate moderate dependence, 91-99 indicate slight dependence, and a score of 100 indicates independence. Higher scores reflect better self-care ability and a higher level of independence.
Psychological health | All participants will undergo an initial measurement within 4 hours of admission, followed by the second and third measurements after the 5-day intervention and on the day of discharge, an average of 11 days, respectively.
  Using the Hospital Anxiety and Depression Scale. This scale focuses on the assessment of emotional symptoms and consists of 14 items, including 7 items for anxiety and 7 items for depression. It uses a four-point Likert-type scoring system, with some items reverse scored. The total score ranges from 0 to 42, with the anxiety subscale ranging from 0 to 21 and the depression subscale ranging from 0 to 21. Higher scores indicate more pronounced anxiety or depressive symptoms. Subscale scores of ≤7 indicate no anxiety or depression, scores of 8-10 indicate possible anxiety or depression, and scores of ≥11 indicate the presence of anxiety or depression.

CONTACTS AND LOCATIONS:
Locations (1):
- TriServiceGH, Taipei, Neihu Dist, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol